CLINICAL TRIAL: NCT05205070
Title: A Phase 2, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Efficacy and Safety of Rosnilimab (ANB030) in the Treatment of Subjects With Alopecia Areata
Brief Title: A Study to Evaluate the Efficacy and Safety of Rosnilimab (ANB030) in Treatment of Subjects With Moderate-to-Severe Alopecia Areata
Acronym: AZURE
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: AnaptysBio, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ANB030-201
Record Dates: First submitted 2022-01-11; First posted 2022-01-24 (Actual); Last update posted 2022-05-10 (Actual); Status verified 2022-05

CONDITIONS: Alopecia Areata
Keywords: PD-1 receptor; Rosnilimab
MeSH Terms: conditions — Alopecia Areata

STUDY DESIGN:
Intervention Model Description: Double-blinded, Placebo controlled, 2:1 ratio of Investigational Product vs Placebo
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blinded design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Rosnilimab (ANB030) (Experimental): ANB030 biological humanized monoclonal antibody, SC injections every 4 weeks
  Interventions: Biological: Rosnilimab
- Placebo solution (Placebo Comparator): Placebo solution, SC injections every 4 weeks
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Rosnilimab — humanized monoclonal antibody
  Other Names: ANB030
  Arms: Rosnilimab (ANB030)
Biological: Placebo — Placebo solution
  Arms: Placebo solution

SUMMARY:
Efficacy and safety of rosnilimab (ANB030) in subjects with moderate-to-severe Alopecia Areata

DETAILED DESCRIPTION:
This is a Phase 2, randomized, double-blind, placebo-controlled, parallel-group,multicenter study to evaluate the safety, tolerability, and efficacy of rosnilimab in subjects with alopecia areata (AA).This study also will evaluate the pharmacokinetics (PK) and pharmacodynamics (PD) of rosnilimab and evaluate the immunogenicity of rosnilimab in subjects with AA.

ELIGIBILITY:
Inclusion Criteria:

* Male or nonpregnant, nonlactating female subject aged 18 to 75 years (inclusive) at the time of informed consent.
* Subjects with a clinical diagnosis of AA defined as having a SALT score ≥ 50 and in which the current episode of hair loss is > 24 weeks (without evidence of spontaneous terminal hair regrowth ≥ 10% within 24 weeks at the time of screening and baseline), but ≤ 8 years (from onset of current episode).

Exclusion Criteria:

* Concomitant active systemic diseases (except stable thyroid diseases) that may cause hair loss (eg, lupus erythematosus, systemic sclerosis, celiac disease) that could interfere with the Investigators' ability to evaluate the subject's response to therapy.
* Subject's cause of hair loss is indeterminable and/or in addition to AA they have concomitant causes of alopecia, such as traction alopecia, cicatricial alopecia, lichen planopilaris, frontal fibrosing alopecia, advanced androgenetic alopecia (ie, Ludwig Type III or Norwood-Hamilton Stage ≥ V), telogen effluvium, trichotillomania, or diffuse AA (alopecia areata incognita).
* Known or suspected congenital or acquired immunodeficiency state, or condition that would compromise the subject's immune status (eg, history of splenectomy).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2021-12-22 (Actual); Primary Completion 2023-01-19 (Estimated); Study Completion 2023-03-19 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in Severity of Alopecia Tool (SALT) score at Week 24 | Week 24

CONTACTS AND LOCATIONS:
Overall Officials: Bruce Randazzo, MD, Study Director — AnaptysBio, Inc.
Locations (16):
- United States (16):
  - 10-105, Birmingham, Alabama
  - Site10-103, Encinitas, California
  - Site 10-113, Northridge, California
  - Site 10-115, Chicago, Illinois
  - 10-104, Indianapolis, Indiana
  - Site 10-109, Plainfield, Indiana
  - Site 10-116, Louisville, Kentucky
  - Site 10-117, Clarkston, Michigan
  - Site 10-111, New York, New York
  - Site 10-101, Charlotte, North Carolina
  - Site 10-102, Bexley, Ohio
  - Site 10-106, Tulsa, Oklahoma
  - 10-107, Upper Saint Clair, Pennsylvania
  - 10-110, Houston, Texas
  - Site 10-108, San Antonio, Texas
  - Site 10-114, Kenosha, Wisconsin

IPD SHARING:
Plan to Share IPD: No